CLINICAL TRIAL: NCT07324291
Title: Prospective Cohort Study of Perianal MBL-CRE Colonization and Infection in Allogeneic Hematopoietic Stem Cell Transplant Recipients
Brief Title: Perianal MBL-CRE Colonization and Infection in Allogeneic Hematopoietic Stem Cell Transplant Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QTJC2024065
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION; Carbapenem-resistant Enterobacterales

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens (perianal swab isolates of CRE) will be retained. DNA will be extracted from MBL-CRE isolates for whole-genome sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to characterize the clinical features of metallo-β-lactamase-producing carbapenem-resistant Enterobacterales (MBL-CRE) colonization and subsequent infection in patients after allogeneic hematopoietic stem cell transplantation (HSCT). The study aims to estimate the incidence of perianal MBL-CRE colonization, the proportion of subsequent infections, the associated risk factors, mortality, and the underlying antibiotic resistance mechanisms.

The main questions this study seeks to answer are:

1. What is the incidence of perianal MBL-CRE colonization following allogeneic HSCT?
2. Among colonized patients, what proportion subsequently develop MBL-CRE infections?
3. What are the risk factors for colonization and infection, the patterns of antimicrobial resistance, and the mortality among infected patients? Participants will undergo perianal swab screening for CRE as part of their routine post-transplant care. MBL-CRE isolates identified from perianal swabs will undergo antimicrobial resistance genomic analysis to investigate bacterial transmission dynamics and resistance mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) who received allogeneic hematopoietic stem cell transplantation;

Exclusion Criteria:

* Engraftment failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) who received allogeneic hematopoietic stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of perianal MBL-CRE colonization. | Within 100 days after allogeneic HSCT.
  The proportion of patients who develop perianal colonization with metallo-β-lactamase-producing carbapenem-resistant Enterobacterales (MBL-CRE) following allogeneic hematopoietic stem cell transplantation (HSCT).

SECONDARY OUTCOMES:
Incidence of MBL-CRE Infection Among Colonized Patients. | From the time of colonization to 6 months after HSCT.
  The proportion of patients with documented perianal MBL-CRE colonization who subsequently develop MBL-CRE clinical infection.
Infection-Related Mortality. | 28 days after documented onset of MBL-CRE infection.
  The proportion of patients with MBL-CRE infection who die due to infection-related causes within 28 days after onset of infection.
All-Cause Mortality. | 28 days after documented onset of MBL-CRE infection.
  The proportion of patients with MBL-CRE infection who die from any cause within 28 days after infection onset.
Clinical Cure Rate | 28 days (range: 25-31 days) after initiation of antimicrobial therapy
  The proportion of MBL-CRE-infected patients who achieve complete clinical resolution of infection-related signs and symptoms after treatment.
Microbiological Eradication Rate. | 14 days (range: 11-17 days) and 28 days (range: 25-31 days) after initiation of antimicrobial therapy.
  The proportion of infected patients with documented clearance of MBL-CRE from repeat culture specimens after treatment.
Risk Factors for MBL-CRE Colonization and Infection | From transplantation to 6 months post-transplant.
  Identification of clinical, demographic, and treatment-related variables associated with perianal MBL-CRE colonization and subsequent infection.